CLINICAL TRIAL: NCT02177539
Title: A New More Efficient Cycloplegia Scheme
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-344
Record Dates: First submitted 2014-05-27; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Refractive Errors
Keywords: cycloplegia; refraction in children; cycloplegic agents; cycloplegic schemes; cyclopentolate
MeSH Terms: conditions — Refractive Errors | interventions — Cyclopentolate; Oxymetazoline; Tropicamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclopentolate (Active Comparator)
  Interventions: Drug: Cyclopentolate; Drug: Cyclopentolate+tropicamide+phenylephrine
- Cyclopentolate+tropicamide+phenylephrine (Experimental)
  Interventions: Drug: Cyclopentolate; Drug: Cyclopentolate+tropicamide+phenylephrine

INTERVENTIONS:
Drug: Cyclopentolate — Traditional scheme. Cyclopentolate, repeat dosage 5 minutes and then wait 40 minutes to retinoscopy. Total wait 45 minutes.
  Other Names: Cyclogyl
Drug: Cyclopentolate+tropicamide+phenylephrine — New scheme. All drugs together and wait 30 minutes for retinoscopy
  Other Names: Cyclogyl, Mydfrin, Mydriacyl

SUMMARY:
The purpose of this study is to determine whether tropicamide + phenylephrine cyclopentolate + applied for once waiting 30 minutes to retinoscopy (new scheme) is not inferior to apply cyclopentolate alone and wait 45 minutes to retinoscopy (traditional scheme)

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 and 10 years

Exclusion Criteria:

* Strabismus
* Ocular surgery
* Another ocular disease than ametropias (i.e uveitis, cataract)
* Cardiovascular or neurologic disease.
* Allergy to any of drugs used in the study

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change in Spherical equivalent | average 18 days
  In the first and second visit the spherical equivalent will be measured with retinoscopy.
  Change in spherical equivalent refraction from first visit to day average 18 days (second visit). On both visits the patient will receive different cyclopegia schemes.

SECONDARY OUTCOMES:
Change in spherical refraction | average 18 days
  Change in spherical refraction between visit 1 and 2.
Change in cylindrical refraction | average 18 days
  Change in cylindrical refraction between visit 1 and 2
iris motility | average 18 days
  both schemes are effective in cycloplegia ? In visit 1 and 2 the iris motility after the cyclopegic schemes will be evaluated

OTHER OUTCOMES:
crying with the application | average 18 days
  does the child cry with both schemes?
eyes color and cycloplegia | average 18 days
  there is a difference between the effectiveness of the schemes according to eye color?

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Salgado, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Departamento de Oftalmología, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Fan DS, Rao SK, Ng JS, Yu CB, Lam DS. Comparative study on the safety and efficacy of different cycloplegic agents in children with darkly pigmented irides. Clin Exp Ophthalmol. 2004 Oct;32(5):462-7. doi: 10.1111/j.1442-9071.2004.00863.x. PMID 15498055
- [Background] McMullen M, Netland PA. Wait time as a driver of overall patient satisfaction in an ophthalmology clinic. Clin Ophthalmol. 2013;7:1655-60. doi: 10.2147/OPTH.S49382. Epub 2013 Aug 20. PMID 23986630
- [Background] Bagheri A, Givrad S, Yazdani S, Reza Mohebbi M. Optimal dosage of cyclopentolate 1% for complete cycloplegia: a randomized clinical trial. Eur J Ophthalmol. 2007 May-Jun;17(3):294-300. doi: 10.1177/112067210701700303. PMID 17534806
- [Background] Alimgil ML, Erda N. [The cycloplegic effect of atropine in comparison with the cyclopentolate-tropicamide-phenylephrine combination]. Klin Monbl Augenheilkd. 1992 Jul;201(1):9-11. doi: 10.1055/s-2008-1045860. German. PMID 1513131
- [Background] Ebri A, Kuper H, Wedner S. Cost-effectiveness of cycloplegic agents: results of a randomized controlled trial in nigerian children. Invest Ophthalmol Vis Sci. 2007 Mar;48(3):1025-31. doi: 10.1167/iovs.06-0604. PMID 17325142
- [Background] Manny RE, Fern KD, Zervas HJ, Cline GE, Scott SK, White JM, Pass AF. 1% Cyclopentolate hydrochloride: another look at the time course of cycloplegia using an objective measure of the accommodative response. Optom Vis Sci. 1993 Aug;70(8):651-65. doi: 10.1097/00006324-199308000-00013. PMID 8414387
- [Background] Twelker JD, Mutti DO. Retinoscopy in infants using a near noncycloplegic technique, cycloplegia with tropicamide 1%, and cycloplegia with cyclopentolate 1%. Optom Vis Sci. 2001 Apr;78(4):215-22. doi: 10.1097/00006324-200104000-00010. PMID 11349929
- [Background] Kleinstein RN, Mutti DO, Manny RE, Shin JA, Zadnik K. Cycloplegia in African-American children. Optom Vis Sci. 1999 Feb;76(2):102-7. doi: 10.1097/00006324-199902000-00017. PMID 10082056
- [Background] Jones LW, Hodes DT. Possible allergic reactions to cyclopentolate hydrochloride: case reports with literature review of uses and adverse reactions. Ophthalmic Physiol Opt. 1991 Jan;11(1):16-21. PMID 2034449
- [Background] Rengstorff RH, Doughty CB. Mydriatic and cycloplegic drugs: a review of ocular and systemic complications. Am J Optom Physiol Opt. 1982 Feb;59(2):162-77. PMID 7039329
- [Background] Hofmeister EM, Kaupp SE, Schallhorn SC. Comparison of tropicamide and cyclopentolate for cycloplegic refractions in myopic adult refractive surgery patients. J Cataract Refract Surg. 2005 Apr;31(4):694-700. doi: 10.1016/j.jcrs.2004.10.068. PMID 15899444
- [Background] Egashira SM, Kish LL, Twelker JD, Mutti DO, Zadnik K, Adams AJ. Comparison of cyclopentolate versus tropicamide cycloplegia in children. Optom Vis Sci. 1993 Dec;70(12):1019-26. doi: 10.1097/00006324-199312000-00005. PMID 8115124
- [Background] Chen J, Xie A, Hou L, Su Y, Lu F, Thorn F. Cycloplegic and noncycloplegic refractions of Chinese neonatal infants. Invest Ophthalmol Vis Sci. 2011 Apr 14;52(5):2456-61. doi: 10.1167/iovs.10-5441. PMID 21087952
- [Background] Salazar M, Shimada K, Patil PN. Iris pigmentation and atropine mydriasis. J Pharmacol Exp Ther. 1976 Apr;197(1):79-88. PMID 1263134
- [Background] Nishizawa AR, Orton RB, Cadera W. Comparison of 0.5% cyclopentolate plus 0.5% tropicamide and 1% cyclopentolate alone for mydriasis of dark irides. Can J Ophthalmol. 1988 Dec;23(7):299-300. PMID 3228775
- [Background] Lovasik JV. Pharmacokinetics of topically applied cyclopentolate HCl and tropicamide. Am J Optom Physiol Opt. 1986 Oct;63(10):787-803. doi: 10.1097/00006324-198610000-00001. PMID 3777109
- [Background] Lovasik JV, Kergoat H. Time course of cycloplegia induced by a new phenylephrine-tropicamide combination drug. Optom Vis Sci. 1990 May;67(5):352-8. doi: 10.1097/00006324-199005000-00009. PMID 2367089
- [Background] Anderson HA, Bertrand KC, Manny RE, Hu YS, Fern KD. Comparison of two drug combinations for dilating dark irides. Optom Vis Sci. 2010 Feb;87(2):120-4. doi: 10.1097/OPX.0b013e3181cc8da3. PMID 20035241
- [Background] Lin LL, Shih YF, Hsiao CH, Su TC, Chen CJ, Hung PT. The cycloplegic effects of cyclopentolate and tropicamide on myopic children. J Ocul Pharmacol Ther. 1998 Aug;14(4):331-5. doi: 10.1089/jop.1998.14.331. PMID 9715436